CLINICAL TRIAL: NCT06834867
Title: A Randomized Controlled Trial of a Multi-component Family Intervention to Lower Depression and Address Intimate Partner Violence (MILAP) Among Young Women in Nepal
Brief Title: Multi-component Family Intervention to Lower Depression and Address Intimate Partner Violence in Nepal
Acronym: MILAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Possible (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH); Wheaton College (Other); Women's Rehabilitation Centre (WOREC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MILAPPossible; 1R01MH135376-01 (NIH)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Intimate Partner Violence (IPV); Depression; PTSD - Post Traumatic Stress Disorder
Keywords: Intimate Partner Violence; Depression; Family Intervention; Mental Health; Nepal; MILAP
MeSH Terms: conditions — Depression; Combat Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial (RCT) with a parallel assignment model. A total of 300 triads (n=900), each consisting of a woman, her husband, and her mother-in-law (MIL), will be randomly assigned in a 1:1 ratio to either the control group (n=150 triads) or the intervention group (n=150 triads).
  Note: We have not seen better option than this one in the drop down menu above.
Who Masked: Outcomes Assessor
Masking Description: The research outcome assessors responsible for collecting data from the study participants will be blinded to the allocation status (intervention vs. enhanced usual care) of each participant. This prevents their assessments from being influenced by any potential bias they might hold regarding the effectiveness of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Usual Care (No Intervention): The control arm will receive enhanced usual care. Counselors (who will be trained by the research team) of the Women's Rehabilitation Centre (WOREC) will conduct initial safety assessment for all participants and offer: a) WOREC's IPV rehabilitation service, which includes a women's shelter, safety and protection from the perpetrator, MH counseling, legal support, and health services; b) educational materials on safety, problems caused by continued IPV, written resources for reducing IPV, and an IPV/DV nationwide hotline; c) referral to wraparound services depending on the woman's needs and priorities: legal support, safe house, psychosocial counseling, health services, and livelihood support services; d) refer to the Nepali government's one-stop IPV center at Janakpur Provincial Hospital and Koshi Hospital in Nepal, and inform them of their options (including support for leaving the relationship if they express that wish).
- MILAP Intervention (Experimental): The MILAP intervention, developed through participatory research and two phases of pilot studies, includes 9 sessions over 9 weeks, totaling 11 hours. MILAP will start with the MilDil component, consisting of two weekly sessions (4 hours total) for mother-in-law (MIL) and daughter-in-law (DIL) dyads, focusing on discussing cultural gender norms and establishing allyship between MIL and DIL. These sessions will be followed by two one-hour sessions on brief Behavioral Activation (BA) to address and prevent depression. After the completion of the MilDil component, the husband-wife dyad will engage in four weekly sessions (4 hours) of Behavioral Couples Therapy (BCT), aimed at improving communication, establishing safety and trust, coping strategies, and fostering caring behaviors between partners. The ninth session (1 hour) will include the triad (woman, husband, and MIL) to review all the lessons learned in the full MILAP intervention, and prepare them to address any challenges.
  Interventions: Behavioral: MILAP intervention

INTERVENTIONS:
Behavioral: MILAP intervention — The MILAP intervention, developed through participatory research, includes 9 sessions over 9 weeks, totaling 11 hours. It begins with the MilDil component, consisting of two sessions (4 hours) for MIL-DIL dyads, focusing on discussing cultural gender norms, raising awareness about the negative impact of IPV, establishing allyship between MIL and DIL, and empowering DILs while enhancing MILs' support for DILs' freedom of movement. This is followed by two one-hour sessions on Brief Behavioral Activation (BA) to address and prevent depression, involving MILs for necessary family support. Lastly, the husband-wife dyad will engage in four weekly sessions (4 hours) of Behavioral Couples Therapy (BCT), aimed at improving communication, coping strategies, and fostering caring behaviors between partners.
  Arms: MILAP Intervention

SUMMARY:
Intimate Partner Violence (IPV) is a major public health problem in low- and middle-income countries (LMICs). Globally, an estimated 30% of women report physical or sexual violence by an intimate partner in their lifetime. IPV is a well-established social driver of mental health problems, and doubles the rate of depression and post-traumatic stress disorder (PTSD). Interventions like cognitive behavioral therapy (CBT) can improve depression after women experiencing IPV exit abusive relationships. However, despite ongoing violence, many young women in LMICs are less likely to divorce or separate from their husband. But ongoing IPV severely limits mental health recovery and increases the risks of suicide. Another important factor in many LMICs is that young women often live in extended, multi-generational households, where studies have shown that mother-in-laws (MILs) play a critical role in young married women's autonomy and freedom of movement, substantially affecting her mental health. The pathways via which multiple family members and ongoing IPV affect young women's mental health in LMICs is very poorly understood. There is an urgent need to design and assess interventions that: a) improve mental health and reduce IPV; b) engage husbands and MILs, and not just women experiencing IPV; and c) elucidate pathways via which IPV-related drivers affect mental health.

This study's research team, with over 16 years of experience in Nepal, conducted a pilot study introducing the Multi-component family Intervention to Lower depression and Address intimate Partner violence (MILAP). MILAP, which translates to "unity and reconciliation" in Nepali, showed promise in reducing depression and IPV among families (comprising women, husbands, and mothers-in-law). Based on these favorable results, the investigators now propose a 12-month randomized controlled trial (RCT) to assess the effectiveness of MILAP in addressing depression, IPV, and PTSD among young married women in Nepal. The goal of this RCT is to assess the effectiveness of MILAP, understand mechanisms of change for MILAP's effectiveness, and conduct a cost-effectiveness analysis. The specific aims of this study are:

AIM 1: Conduct a 12-month RCT to assess the effectiveness of MILAP on depression, IPV, and PTSD among young married women in Nepal.

AIM 2: Conduct a mixed-methods assessment of theorized mechanisms of change for MILAP's effectiveness.

AIM 3: Conduct a cost-effectiveness analysis of MILAP for depression and IPV.

Participants of this study will receive either MILAP or enhanced usual care, and will answer questions about depression, IPV and PTSD at baseline, at 1 month and every 3 months until 1-year.

DETAILED DESCRIPTION:
Intimate Partner Violence (IPV), defined as control, psychological, physical, and sexual violence by a close partner, is a major public health problem in low- and middle-income countries (LMICs) with one in three women experiencing IPV in their lifetime. National prevalence in Nepal, this study's research site, is 25% for IPV and 12% for depression. IPV is a well-established driver of mental health (MH) problems, doubling the rate of depression via feelings of worthlessness, disempowerment, amotivation, social isolation and marital strain, and increasing the incidence of post-traumatic stress disorder (PTSD) via trauma, increased fear and anxiety. The association between IPV and MH problems is well- documented in South Asia, with 25-50% of women with IPV reporting depressive symptoms and an increase in rates of PTSD.

Several meta-analyses have highlighted the lack of interventions to reduce IPV and improve MH in LMICs. A major challenge is that despite ongoing IPV, young women in LMICs are less likely to have the ability and/or desire to undergo divorce or separation. This substantially limits the impact of available interventions such as CBT (cognitive behavioral therapy), which has been found to improve depression among women who have already exited relationships that led to IPV. Review articles have thus concluded that there is a significant gap in behavioral interventions that can improve outcomes for women who are currently experiencing abuse. Thus, a culturally appropriate evidence-based intervention is needed to enhance MH recovery while simultaneously reducing IPV.

Many women in LMICs live in multi-generational households, where the drivers of IPV and MH include not just the husband, but often the mother-in-law (MIL). There is evidence that MILs play a substantial role in restricting or supporting the daughter-in-law's (DIL's) Freedom of Movement (FOM), as young women (age 15-24) move into their husband's home. Combined with the evidence that MILs also affect IPV or perpetrate direct violence, they have a critical role in driving or mitigating the complex relationship between IPV and MH. Despite this, majority of IPV and MH interventions involve only the women experiencing IPV, and rarely also their husbands, but not the whole family unit.

This study's investigators developed and pilot-tested a novel Multi-component family Intervention to Lower depression and Address intimate Partner violence (MILAP, meaning unity and reconciliation in Nepali) among young married women in Nepal. MILAP engages three members (triads) of each family, i.e wives (also frequently referred as daughter-in-laws(DILs) throughout the description), and their husbands and MILs. MILAP's first component engages DILs and their MILs by establishing them as allies in addressing IPV and improving DIL's empowerment and freedom of movement. In MILAP's second component, the wife and husband participate in behavioral couples therapy (BCT) to improve communication skills, increase caring behaviors, and enhance trust in the marital relationship. This approach was highly acceptable to the participants as the intervention focused on skills-building and relationships rather than explicitly dealing with the stigmatizing topics of IPV and mental health. The intervention was found to be safe and feasible, and resulted in substantial reduction in proportion of people with moderate depression and frequency of IPV. Based on this pilot study, the investigators now propose to conduct a randomized controlled trial (RCT) of MILAP to establish intervention's effectiveness, understand mechanism of intervention impact, and conduct a costing analysis. Additionally, the investigators aim to understand the processes via which MILAP addresses IPV-related drivers of MH. For this, the investigators will conduct a mixed-methods explanatory assessment of the MILAP's theorized mechanisms of change by combining data from quantitative and qualitative assessments. Finally, the investigators will conduct a cost-effectiveness analysis of MILAP for depression and IPV to estimate the health and economic benefits of investing in delivering MILAP. This analysis will use programmatic and financial data to perform a comprehensive analysis of costs incurred in providing MILAP. The purpose of this analysis is to assist policymakers/payors in assessing MILAP for potential investment by providing: a) assessment of average costs to deliver MILAP for each family (triad); b) estimation of incremental average costs for MILAP over enhanced usual care per family (triad); and c) disaggregation of costs in delivering MILAP's components (MilDil and BCT).

This study will include family units (triads) which will be randomized 1:1 to the intervention group and control group. The study will involve 900 participants from 300 triads (wife, her husband and MIL) where 150 triads will be assigned to intervention group and 150 triads will be assigned to control group. The mobilized community health workers (CHWs) will refer potential candidates from the community to recruitment sites where the staffs will screen the referred individuals for eligibility. Research staff trained by investigators will conduct initial screening for presence of IPV using a screening tool adapted from International Violence Against Women Survey (IVAWS). Initial screening will be made in community-based organizations and women's groups, which are well-attended and hosted by our community-based partner organization, Women's Rehabilitation Centre (WOREC)'s offices. If the woman (wife) meets the criteria, she will be asked to provide permission for the research team to approach her husband and MIL about participating in the study. If her response is positive, she will be asked to choose the most appropriate way to engage her husband and MIL: a) she will bring them to the next visit; or b) the research staff will call them directly and ask them to come to the recruitment location; or c) the CHWs will approach the husband and MIL at their home. After verbal consent with all three members of the family (consent will be obtained from each member separately), the research staff will engage participants in the written informed consent process, which will also happen individually for each of the 3 family members. After the consent process, the research staff will conduct baseline assessments with the wive, husband and MIL participants separately. Then, the research staff will randomly assign the triads to intervention or control arm. Prior to the start of the intervention, a statistician not directly involved with the implementation of the study will draw up a computer generated "random order of assignment" list. These random assignments will be placed in advance in sealed, numbered envelopes, so research staff is not aware of the upcoming assignment. At the end of the baseline assessment session, the randomization assignment will be revealed to the triad by drawing the next available envelope in their presence. Assessment staff will be blinded from allocation status. Enhanced usual care will be delivered by WOREC-based counselors (called "psychosocial counselors", and widely available in Nepal) who will not be trained in intervention components. The intervention i.e. MILAP will be delivered by research counselors, who will be trained and supported by the research team.

Blinded research staff will conduct assessments at baseline (after obtaining consent), at 1 month (between MilDil and BCT) and every 3 months until 1-year follow-up. Based on the pilot studies, the investigators estimate that assessments will last between 45-75 minutes (longer for the wives as they will complete more assessments). Research staff will collect contact information at baseline and update it at follow-ups. Staff will receive training and certification on interviewing and assessments, strategies to reduce social desirability bias, avoid questions that may reveal if the participant is in the intervention or control arm, and follow human subjects protections and the study protocol. All assessments will be conducted in local languages and in a private room at the WOREC's office, or at a different mutually convenient location that provides privacy. Responses will be entered into a tablet-based version of Research Electronic Data Capture (REDCap). This study will use following tools to collect data from participants:

1. Demographic Information - Age, education, languages spoken, religion, income, caste, migrant status, marital status and number of months since wedding date
2. Adverse Childhood Experiences: 8 items each on witnessing and experiencing adverse childhood events. For MIL, additional questions from IVAWS on history of experiencing IPV
3. Patient Health Questionnaire-9 (PHQ-9): 9-items scale to measure depression among women participants
4. Indian Family Violence and Control Scale (IFVCS): 63-items tool to measure abusive control, psychological, physical and sexual violence perpetrated by an intimate partner
5. Post Traumatic Stress Disorder (PTSD) Checklist -Civilian Version (PCL-C): 17-itemed self-report rating scale for PTSD
6. Women's Autonomy Scale: 5 itemed tool to measure women's ability to move outside the household unescorted
7. Gender Equitable Men Scale (GEMS): 4-item, 3-point response subscale pertaining to IPV
8. Anxiety Sensitivity Scale (ASI): 16 items to assess perceived threat level
9. Fear Survey Schedule (FSS): Subscale for injury and sex aggression fears
10. Spousal Quality Relationship Scale (SQRS): 21 items on commitment, trust and satisfaction between partners; MILRQS: 7 items on MIL-DIL relationship
11. Behavioural Activation and Depression Scale - Short Form (BADS-SF): 9 items to assess withdrawal from or engagement in rewarding activities
12. Rosenberg Self Esteem Scale (RSES): 10 items to globally self-worth by measuring positive and negative feelings about self
13. Sexual Relationship Power Scale (SRPS): 8 items subscale for decision making power in the relationship
14. World Health Organization Quality of Life-BREF (WHOQOL-BREF): 9 items on psychological well-being and social functioning
15. World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0): 16-item tool to measure health and disability across cultures.
16. General Anxiety Disorder (GAD-7): 7 items to screen generalized anxiety disorder

Qualitative data will be collected twice from ~15% (n=66 participants based on the resource availability and expected number to reach thematic saturation at 22 triads) of the intervention arm sample, through serial in-depth interviews (IDIs). Triads will be purposively selected based on variation in engagement with MILAP intervention activities. All IDIs will follow a semi-structured guide and will be implemented by experienced staff members fluent in local languages and trained in safety and response procedures. Serial IDIs will be conducted at two timepoints: at the end of MILAP intervention and at the 12-month follow up visit.

The effectiveness of MILAP to reduce the proportion of women (DILs) with moderate to severe depression (primary outcome), levels of IPV (primary outcome), and PTSD (secondary outcomes) significantly more than enhanced usual care will be assessed via intention-to-treat (ITT) regression analyses at the end of the trial (12-month follow-up, a single timepoint), as well as longitudinally via the interaction between intervention arm and time in a two-level regression model with repeated measures nested within participants (=DIL) and a random intercept for participants. This will be a logistic regression model for the binary depression outcome, and a linear model for the continuous IPV (IFVCS score) and PTSD (PCL-C score) outcomes.

The investigators will conduct a mixed-methods explanatory assessment of the intervention's theorized mechanisms of change by combining data from the full cohort of quantitative assessments and from serial IDIs with 22 families to understand the processes via which the intervention addresses IPV-related drivers of MH. Analyses of the IDI transcripts will use a thematic approach to coding and summarization using Dedoose qualitative data analysis software. A preliminary codebook will be developed from interview guides and rapid analysis content, then refined after all analysts code a set of transcripts independently and resolve discrepancies through consensus. The remaining transcripts will be single-coded, maintaining intercoder reliability of at least 80% throughout the coding process using coding test features of Dedoose and subsequent kappa calculations. Coding memos will be used to summarize and explore the relationship between the constructs of the theory of change framework (e.g., the relationship between intervention processes and hypothesized mechanisms of change, or between mechanisms of change and outcomes, allowing triangulation with quantitative data). Analysts will also review and analyze coded serial IDI content within each participant's dataset to look specifically for patterns over time to further understand sustained results. Findings from the qualitative and quantitative analyses will be triangulated to build a more comprehensive understanding of how the hypothesized changes in mechanisms of action resulted in the intended outcomes and their relative weight in creating change. Both differences and similarities in the sets of data will be examined and presented to understand the relationship between the constructs in the conceptual model and to highlight any factors that may be uniquely identified by qualitative or quantitative methods. These data will inform interpretation of the effectiveness findings and next steps for any refinements that may be necessary for scale-up.

The cost-effectiveness analysis will be performed using programmatic and financial data for the duration of delivering intervention. The costs measured will include: a) MILAP intervention costs, b) enhanced usual care costs, and c) informal service sector costs. The analysis will use bottom-up or micro-costing approach at the beneficiary (triad) level to estimate the MILAP intervention costs. These costs will include direct and indirect facility-level costs that are recurrent and are related to depreciation and/or amortization of capital cost. Total cost at the facility per beneficiary will be calculated, and through repeated measurements the average facility-level MILAP intervention costs will be estimated. Our primary approach for analyzing facility-level MILAP costs is Time Defined Activity Based Costing (TDABC), a beneficiary-centered costing method that studies resources use in delivering services and measures detailed resource use throughout service delivery. Costs of enhanced usual care will include costs of a counselor, IPV rehabilitation service, education materials, and costs of referral to wraparound services and referral to one-stop IPV center at provincial hospitals, as applicable. Informal service sector costs will include beneficiary (triad) time costs, transportation costs, and other intervention-specific costs that are borne by the beneficiary (triad) in either MILAP intervention or enhanced usual care group. At the completion of comprehensive costing, the investigators will evaluate the difference in outcomes of interest in the MILAP intervention group compared to the enhanced usual care group, and estimate the incremental costs per difference in unit outcome. The service systems reference case only includes formal service sector costs in MILAP or enhanced care. The investigators will collect both programmatic and financial data during the implementation period using the following sources: a) time inputs of counselors in delivering MILAP recorded as time stamps in routine logs, b) financial data on non-counselor costs, c) program records and financial data on costs incurred in enhanced usual care, and d) survey inputs from participants on informal service sector costs at baseline, intermediate, and end-line surveys. The outcome data are extracted from program records.

If successful, this study will provide the governments of Nepal and other LMICs with an integrated intervention and a set of implementation strategies to deliver interventions for reducing proportion of women reporting moderate to severe depression and IPV.

ELIGIBILITY:
Inclusion Criteria:

* Married women aged 15-24 years, their husbands and MILs sharing a household;
* Living in the catchment area with no stated intention of leaving during the study period;
* Participants speaking in Maithili or Nepali;
* Wife reporting Intimate Partner Violence (physical, sexual or abusive control) in last 12 months as measured by three questions from the International Violence Against Women Survey (IVAWS);
* Expressing desire to remain in the current relationship/family

Exclusion Criteria:

* Pregnant women;
* History of IPV severe enough to result in hospitalization in the past 12 months;
* Significant cognitive problems/disability precluding participation;
* Any participant with Severe Alcohol Dependence, defined as Severity of Alcohol Dependence Questionnaire (SADQ) > 31 (those with mild to moderate dependance will be referred but not excluded)

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who have moderate to severe depression | Assessments at baseline, and at 1, 3, 6, 9 and 12 months follow-ups.
  Patient Health Questionnaire (PHQ-9) is a widely used instrument for screening, diagnosing, and monitoring the severity of depression. It consists of 9 items, each scored from 0 (not at all) to 3 (nearly every day), with a total possible score ranging from 0 to 27. Higher scores reflect greater severity of depressive symptoms, making the PHQ-9 a valuable tool for assessing the impact of interventions on depression levels. This study will use PHQ-9 score as continuous variable and assess proportion of women whose PHQ-9 score is greater than 9 at 12-month follow-up
Abusive control, physical violence, and sexual violence/coercion | Assessment at baseline, and at 1, 3, 6, 9, and 12 months follow-ups
  This study will measure abusive control, physical violence, and sexual violence/coercion using the Indian Family Violence and Control Scale (IFVCS), which is specifically designed to assess and quantify various forms of violence and controlling behaviors within family contexts. It includes 75 items on physical, emotional, and financial abuse, along with behaviors aimed at exerting control, particularly within marital relationships. This study will use 63 items, out of total 75 items, that are relevant to the study outcomes. Higher score explains high control and violence over women. The score ranges from 14 to 56.

SECONDARY OUTCOMES:
Post-traumatic Stress Disorder (PTSD) Symptom Severity | Assessments at baseline, and at 1, 3, 6, 9, and 12 months follow-ups.
  This study will assess post-traumatic stress disorder (PTSD) symptom severity using the PTSD Checklist - Civilian Version (PCL-C). It is a 17-items self-rated measure that assesses PTSD symptom severity based on the DSM-4 PTSD criteria. The score ranges from 17 to 85. Higher score explains higher level of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Bibhav Acharya, MD, Principal Investigator — University of California, San Francisco; Sabitri Sapkota, PhD, Principal Investigator — Possible
Locations (1):
- Possible, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified quantitative data collected using our qualitative tools, including NIH's Common Data Elements relevant to our study . For qualitative data, we will share the structured notes.
Supporting Information: SAP, Analytic Code
Time Frame: IPD and supporting information will be available approximately 12 months following the end of the trial (April 1, 2030). IPD will be available to the research community in perpetuity.
Access Criteria: All shared data will be publicly accessible in the National Institute of Mental Health (NIMH) Data Archive (NDA).
URL: https://nda.nih.gov/;https://nda.nih.gov/nda/nimh-common-data-elements

REFERENCES:
- [Background] Sapkota D, Baird K, Saito A, Anderson D. Interventions for reducing and/or controlling domestic violence among pregnant women in low- and middle-income countries: a systematic review. Syst Rev. 2019 Apr 2;8(1):79. doi: 10.1186/s13643-019-0998-4. PMID 30940204
- [Background] Bean J, Moller AT. Posttraumatic stress and depressive symptomatology in a sample of battered women from South Africa. Psychol Rep. 2002 Jun;90(3 Pt 1):750-2. doi: 10.2466/pr0.2002.90.3.750. PMID 12090502
- [Background] Marahatta K, Samuel R, Sharma P, Dixit L, Shrestha BR. Suicide burden and prevention in Nepal: The need for a national strategy. WHO South East Asia J Public Health. 2017 Apr;6(1):45-49. doi: 10.4103/2224-3151.206164. PMID 28597859
- [Background] Rimal P, Choudhury N, Agrawal P, Basnet M, Bohara B, Citrin D, Dhungana SK, Gauchan B, Gupta P, Gupta TK, Halliday S, Kadayat B, Mahar R, Maru D, Nguyen V, Poudel S, Raut A, Rawal J, Sapkota S, Schwarz D, Schwarz R, Shrestha S, Swar S, Thapa A, Thapa P, White R, Acharya B. Collaborative care model for depression in rural Nepal: a mixed-methods implementation research study. BMJ Open. 2021 Aug 16;11(8):e048481. doi: 10.1136/bmjopen-2020-048481. PMID 34400456
- [Background] Patel AR, Prabhu S, Sciarrino NA, Presseau C, Smith NB, Rozek DC. Gender-based violence and suicidal ideation among Indian women from slums: An examination of direct and indirect effects of depression, anxiety, and PTSD symptoms. Psychol Trauma. 2021 Sep;13(6):694-702. doi: 10.1037/tra0000998. Epub 2021 Jan 28. PMID 33507794
- [Derived] Shrestha M, Heylen E, Sigdel K, Dhimal M, Nepal P, Pant P, Jha RK, Rimal R, Khatri R, Joshi S, Sharma S, Shrestha S, Poudel S, Mainali S, Sapkota S, Acharya B. A randomized controlled trial of a multi-component family intervention to lower depression and address intimate partner violence (MILAP) among young married women in Nepal: a study protocol. Res Sq [Preprint]. 2025 Sep 9:rs.3.rs-7048952. doi: 10.21203/rs.3.rs-7048952/v1. PMID 40964025